CLINICAL TRIAL: NCT07128849
Title: Effects of Phase I Cardiac Rehabilitation With and Without Upper Limb Cycle Ergometer in Immediate Post-Operative Period of CABG
Brief Title: Effect of Phase I Cardiac Rehab With or Without Upper Limb Cycle Ergometer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/RCR & AHS/24/0351
Record Dates: First submitted 2025-07-21; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: CAD
Keywords: phase I cardiac rehabilitation; upper limb cycle ergometer; post op period CABG

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- upper limb exercise with arm ergometer (Experimental): Group A will receive upper limb exercise on arm ergometer lasting 5 min at 30 rpm (Rotation per minute) 3 times a day for 7 days and standard treatment which includes breathing exercises (3 sets of 10 repetitions daily for 7 days); active upper and lower exercises (3 sets of 10 repetitions daily for 7 days) with bed inclined at 45°; ambulation within the inpatient wards for 6 min, transfer to chair (allocated at the side of bed sitting for 30min), that will be progressed as patient condition till 7th day
  Interventions: Other: upper limb exercise with arm ergometer
- upper limb exercise with out arm ergometer (Active Comparator): Group B will receive standard treatment which includes breathing exercises (3 sets of 10 repetitions daily for 7 days); active upper and lower exercises (3 sets of 10 repetitions daily for 7 days) with bed inclined at 45°; ambulation within the inpatient wards for 6 min, transfer to chair (allocated at the side of bed sitting for 30min), that will be progressed as patient condition till 7th day
  Interventions: Other: upper limb exercise with out arm ergometer

INTERVENTIONS:
Other: upper limb exercise with arm ergometer — upper limb exercise on arm ergometer lasting 5 min at 30 rpm (Rotation per minute) 3 times a day for 7 days and standard treatment which includes breathing exercises (3 sets of 10 repetitions daily for 7 days); active upper and lower exercises (3 sets of 10 repetitions daily for 7 days) with bed inclined at 45°; ambulation within the inpatient wards for 6 min, transfer to chair (allocated at the side of bed sitting for 30min), that will be progressed as patient condition till 7th day
  Arms: upper limb exercise with arm ergometer
Other: upper limb exercise with out arm ergometer — standard treatment which includes breathing exercises (3 sets of 10 repetitions daily for 7 days); active upper and lower exercises (3 sets of 10 repetitions daily for 7 days) with bed inclined at 45°; ambulation within the inpatient wards for 6 min, transfer to chair (allocated at the side of bed sitting for 30min), that will be progressed as patient condition till 7th day
  Arms: upper limb exercise with out arm ergometer

SUMMARY:
The aim of the study is to investigate the effects of an upper limb cycle ergometer in phase I CABG patients. This will likely enhance various outcomes such as quality of life, dyspnea, functional outcome measure, cardiovascular parameters, and upper limb mobility. If utilized, the arm ergometer may contribute to improve upper limb strength and endurance. This could result in improving upper limb range of motion and reducing the risk of adhesive capsulitis. This study will positively impact society by reducing morbidity and mortality rates, healthcare costs and ultimately improves patient care.

DETAILED DESCRIPTION:
The most often done major surgical surgery is coronary artery bypass grafting (CABG), a significant surgical procedure by using harvested venous or arterial conduit to bypass atheromatous obstructions in a patient's coronary arteries. Following heart surgery, patients face many complications that increases the duration of stay in the intensive care unit (ICU) and hospital, as well as the death rates following surgery. Following coronary artery bypass grafting (CABG), compliance with the cardiac rehabilitation (CR) regimen is essential. Cardiac rehabilitation in phase I include mobilization, respiratory and physical exercises, education on heart disease risk factors, and stress and anxiety management. An apparatus designed to help physiotherapists to increase muscle training is the upper limb cycle ergometer. It is possible to execute cyclical rotations with this equipment and utilize it for resistive, active, and passive patient exercise. Patients who have had coronary artery bypass surgery report improved physical and psychosocial functioning after engaging in arm ergometer workouts. The aim of this study is to investigate the effects of phase I cardiac rehabilitation on quality of life, dyspnea, functional outcome measure and cardiovascular parameters with and without upper limb cycle ergometer in immediate post-operative period of CABG.

A randomized clinical trial will be conducted at Combined Military Hospital Lahore. Non-probability convenient sampling technique will be applied on the patients according to the inclusion criteria. Patient will be randomly allocated through lottery method into group A and group B to collect data. Group A will receive upper limb exercise on arm ergometer lasting 5 min at 30 rpm (rotation per minute) 3 times a day for 7 days and standard treatment which includes breathing exercises, active upper and lower exercises (3 sets of 10 repetitions daily for 7 days); ambulation within the inpatient wards for 6 min, transfer to chair (allocated at the side of bed sitting for 30 min), that will be progressed as patient condition till 7th day. Group B will receive same standard treatment as above, but without arm ergometer. The study will be completed within the time duration of ten months. Treatment evaluation of patients will be done after one week through 36-Item Short Form Survey (SF-36), Modified Medical Research Council Dyspnea scale, and Functional Independence Measure scale. Data will be analyzed using SPSS software version 27. After assessing normality of data by Shapiro-wilk test, it will be decided either parametric or non-parametric test will be used within a group or between two groups.

ELIGIBILITY:
Inclusion Criteria:

* Planned CABG patients
* 40-65 years
* Both male and female
* Hemodynamic stable patients
* Post extubation

Exclusion Criteria:

* Patients suffering from pulmonary diseases and thyroid disorders
* Mechanical ventilation more than 24 hr
* Mean arterial pressure i.e, < 60 mmHg or > 140 mmHg and heart rate not more than 120bpm
* Having an orthopedic condition that makes the use of upper and lower extremity impossible.
* Who have neurological impairment influencing breathing rate and heart rate.
* Who required the implantation of an intra-aortic balloon during surgery
* Who experienced postoperative complications such as pulmonary embolism

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-07-17 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Functional independence Measure (FIM) | 7 days
  There are eighteen items in the FIM, and each item has a maximum score of seven points, a minimum score of one point, and and a maximum score of 126 points overall. The FIM has eighteen items, of which thirteen are used to test motor ADL (six self-care items, two sphincter control tasks, three transfer items, and two motor items), and the other five are used to assess cognitive ADL (two items for communication and three items for social cognition).
36- Item Short Form Survey Instrument | 7 days
  The SF-36 brief survey, which includes 36 items across eight categories of QOL, is a standardised tool for assessing generic health concepts. It includes ten items related to physical functioning, four items related to physical problems, five items related to general mental health, three items related to emotional problems, and two items related to relationships with family and friends. General health, which includes six items regarding the patient's personal opinion of health; physical pain, which includes 2 items about the patient's body pain intensity; and energy or vitality, which includes four things about vitality, exhaustion, and tiredness. There are total 8 domains of SF-36 and its score range is from 0-100, the lower score means more disability and higher score means less disability
Modified Medical Research Council (MMRC) Dyspnea Scale | 7 days
  During activity, the 5-item MMRC dyspnea scale was used to measure the severity of dyspnea. On this scale, the degree of dyspnea is rated from 0 (no dyspnea during ordinary activities or vigorous exercise) to 4 (dyspnea during routine activities). The patients were instructed to identify the number on the scale that most accurately represented their dyspnea after reading the descriptive comments. The reliability of the MMRC scale was computed with an intra-class correlation coefficient of 0.8, and the validity of the scale was thus established by using the perspectives of heart, lung, and nursing specialists through the use of the facial and qualitative content validity methodologies

SECONDARY OUTCOMES:
Heart Rate (HR) | 7 days
  Cardiac monitors in ICU/CCU settings will be used to measure heart rate (HR).
Respiratory Rate (RR) | 7 Days
  Cardiac monitors in ICU/ CCU will be used to measure respiratory rate (RR).
Blood Pressure (BP) | 7 Days
  Cardiac monitors in ICU / CCU will be used to measure blood pressure (B.P).
Oxygen Saturation | 7 Days
  Cardiac monitors in ICU / CCU will be used to measure Oxygen saturation.

CONTACTS AND LOCATIONS:
Overall Officials: Iram Nawaz, Mphill, Principal Investigator — Riphah International University
Locations (1):
- Gulab Devi Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Organization WH. Cardiovascular diseases (CVDs). 2021.
- [Background] Bachar BJ, Manna B. Coronary Artery Bypass Graft. 2023 Aug 8. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK507836/ PMID 29939613
- [Background] Alexander JH, Smith PK. Coronary-Artery Bypass Grafting. N Engl J Med. 2016 Sep 8;375(10):e22. doi: 10.1056/NEJMc1608042. No abstract available. PMID 27602683
- [Background] Dimopoulos S, Raidou V, Elaiopoulos D, Chatzivasiloglou F, Markantonaki D, Lyberopoulou E, Vasileiadis I, Marathias K, Nanas S, Karabinis A. Sonographic muscle mass assessment in patients after cardiac surgery. World J Cardiol. 2020 Jul 26;12(7):351-361. doi: 10.4330/wjc.v12.i7.351. PMID 32843937
- [Background] Cordeiro ALL, Mascarenhas HC, Landerson L, Araujo JDS, Borges DL, Melo TA, Guimaraes A, Petto J. Inspiratory Muscle Training Based on Anaerobic Threshold on the Functional Capacity of Patients After Coronary Artery Bypass Grafting: Clinical Trial. Braz J Cardiovasc Surg. 2020 Dec 1;35(6):942-949. doi: 10.21470/1678-9741-2019-0448. PMID 33113311
- [Background] Hossein Pour AH, Gholami M, Saki M, Birjandi M. The effect of inspiratory muscle training on fatigue and dyspnea in patients with heart failure: A randomized, controlled trial. Jpn J Nurs Sci. 2020 Apr;17(2):e12290. doi: 10.1111/jjns.12290. Epub 2019 Aug 19. PMID 31429207